CLINICAL TRIAL: NCT04793204
Title: Pharmacokinetic Study of Fezolinetant - An Open-Label, Single and Multiple Dose Study to Evaluate the Pharmacokinetics and Safety of Fezolinetant in Healthy Chinese Female Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of Fezolinetant in Healthy Chinese Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma China, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2693-CL-0030
Record Dates: First submitted 2021-03-09; First posted 2021-03-11 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
Keywords: Fezolinetant; Pharmacokinetics; ESN364; Healthy Volunteer
MeSH Terms: interventions — fezolinetant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fezolinetant (Experimental): A single oral dose of fezolinetant will be administered with water under fasting conditions on day 1 (low dose), day 4 (medium dose) and day 7 (high dose). From day 10 to day 15, the medium dose of fezolinetant will be administered with water after breakfast once daily. On day 16, the medium dose of fezolinetant will be administered with water under fasting conditions.
  Interventions: Drug: fezolinetant

INTERVENTIONS:
Drug: fezolinetant — oral
  Other Names: ESN364

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of fezolinetant after single-dose and multiple dose administration in healthy Chinese female participants.

DETAILED DESCRIPTION:
Participants will undergo screening evaluations to determine their eligibility within 21 days prior to the study enrollment.

Participants will be admitted to the clinical unit a day before administration (day -1) and will be confined in the clinical unit until 48 hours after last administration (day 18).

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) range of > 19 kg/m^2 and ≤ 24.9 kg/m^2.
* Subject has a body weight at screening ≥ 45.0 kg.
* Subject must either:

  * Be of nonchildbearing potential: Postmenopausal (defined as at least 1 year without any menses for which there is no other obvious pathological or physiological cause) prior to screening, or documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy)
  * Or, if of childbearing potential, agree not to try to become pregnant during the study and for 30 days after the final study drug administration; and have a negative pregnancy test at screening and day -1; and if heterosexually active, agree to consistently use 1 form of effective birth control starting at screening and throughout the study period and for 30 days after the final study drug administration. If male partner has undergone effective surgical sterilization (vasectomy or bilateral orchiectomy), it is not necessary to implement the birth control method.
* Subject must agree not to breastfeed starting at screening and throughout the study period, and for 30 days after the final study drug administration.
* Subject must not donate ova starting at screening and throughout the study period, and for 30 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present study, defined as 84 days prior to the screening test until completion of the last study visit.

Exclusion Criteria:

* Subject has been pregnant within 6 months (including delivery or abortion) or has been breast feeding within 3 months prior to the screening test.
* Subject has had previous exposure with fezolinetant.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema, or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies) prior to study drug administration.
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma-glutamyl transferase [GGT] and total bilirubin [TBL]) above the upper limit of normal at screening or day -1. In such a case, the assessment is allowed to repeated only once.
* Subject applies to any of the following concerns with regard to tuberculosis.

  * History of active tuberculosis
  * Significant abnormalities detected in a chest X-ray test at Screening
  * Contact with infectious tuberculous patients
* Subject had clinically significant abnormality in their laboratory value at screening test and on day -1.
* Subject who deviated from the following range of vital signs or routine 12-lead electrocardiogram (ECG) results at screening test or day -1. If QT interval corrected by Fridericia method (QTcF) exceeds the limits determined, ECG is allowed to be repeated once; if pulse rate or ear temperature exceeds the limits determined, the measurements of pulse and ear temperature are allowed to be repeated once; if the blood pressure exceed limits determined, the measurement of blood pressure should be repeated once. The final judgment should be based on the retest results.
* Subject has a positive serology test for hepatitis B surface antigen (HBsAg), hepatitis B core (HBc) antibody, hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibody, syphilis and hepatitis A virus (HAV) antibodies (immunoglobulin M [IgM]) at screening.
* Subject has used any drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, tricyclic antidepressants, phencyclidine, cocaine and opiates) within 3 months prior to day -1. Subject who has a history of drug abuse within 2 years prior to screening test.
* Subject has used any prescribed or nonprescribed drugs (including vitamins, oral contraceptives, hormone replacement therapy [HRT], natural and herbal remedies, e.g. St. John's Wort, Chinese medicine such as Heyan Kuntai Capsule) in 3 months prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day) and topical dermatological products, including corticosteroid products.
* Subject has used any inducer of metabolism (e.g. barbiturates, rifampin) in 3 months prior to day -1.
* Subject has a history of smoking within 3 months prior to day -1.
* Subject whose daily caffeine consumption is ≥ 500 mg (500 mg of caffeine: about 800 mL of coffee, 1600 mL of black tea, 2500 mL of green tea, 5000 mL of cola).
* Subject whose weekly alcohol consumption is ≥14 units* within 6 months prior to screening test, or who has a history of alcohol dependency, drug dependency, chemical dependency, or alcohol abuse within 2 years prior to screening test (*1 unit: approximately 360 mL of beer, 120 mL of wine, 30 mL of spirit).
* Subject who has had blood sampled or donated blood during the following period.

  * Whole blood sample of ≥ 400 mL: from 90 days prior to screening test until hospital admission.
  * Whole blood sample of ≥ 200 mL: from 30 days prior to screening test until hospital admission.
  * Blood component donation: from 14 days prior to screening test until hospital admission.
* Subject is employed by the sponsor, contract research organization (CRO), or study center associated with this study.
* Subject is deemed unsuitable for participating in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Up to day 41
  Adverse events (AEs) will be coded using medical dictionary for regulatory activities (MedDRA). An AE is any untoward medical occurrence in a participant administered a study drug and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medical product whether or not considered related to the medical product. An AE is considered "serious" if, in the view of either the investigator or sponsor, the event: results in death, is life-threatening, results in persistent or significant disability/incapacity or substantial disruption of the ability to conduct normal life functions, results in congenital anomaly or birth defect, requires hospitalization or prolongation to hospitalization, or other medically important event.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to day 41
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) | Up to day 41
  Number of participants with potentially clinically significant vital sign values.
Number of participants with rountine 12 lead electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) | Up to day 41
  Number of participants with potentially clinically significant ECG values.
Pharmacokinetics (PK) of fezolinetant in plasma: AUC24 | Up to day 7
  Area under the concentration-time curve from the time of dosing to 24 hours (AUC24) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: AUCinf | Up to day 7
  AUC from the time of dosing extrapolated to time infinity (AUCinf) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: AUCinf(%extrap) | Up to day 7
  Percentage of extrapolated section of AUCinf (AUCinf(%extrap)) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: AUClast | Up to day 7
  Area under the concentration time curve from the time of dosing to the last measurable concentration (AUClast) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Ctrough | Up to day 16
  Concentration immediately prior to dosing at multiple dosing (trough concentration) (Ctrough) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: AUCtau | Up to day 16
  AUC from the time of dosing to the start of the next dosing interval (AUCtau) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: CL/F | Up to day 16
  Apparent total clearance after extra-vascular dosing (CL/F) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Cmax | Up to day 16
  Maximum concentration (Cmax) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: PTR | Up to day 16
  Peak-trough ratio (PTR) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Rac(AUC) | Up to day 16
  Accumulation ratio calculated using AUC (Rac(AUC)) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Rac(Cmax) | Up to day 16
  Accumulation ratio calculated using Cmax (Rac(Cmax)) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: t1/2 | Up to day 16
  Terminal elimination half-life (t1/2) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: tmax | Up to day 16
  Time of the maximum concentration (tmax) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Vz/F | Up to day 16
  Apparent volume of distribution during the terminal elimination phase after extra-vascular dosing (Vz/F) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of fezolinetant in plasma: Tlag | Up to day 16
  Time-lag (Tlag) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: AUC24 | Up to day 7
  Area under the concentration-time curve from the time of dosing to 24 hours (AUC24) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: AUCinf | Up to day 7
  Area under the concentration time curve from the time of dosing extrapolated to time infinity (AUCinf) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: AUCinf(%extrap) | Up to day 7
  Percentage of extrapolated section of AUCinf (AUCinf(%extrap)) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: AUClast | Up to day 7
  Area under the concentration time curve from the time of dosing to the last measurable concentration (AUClast) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: Ctrough | Up to day 16
  Concentration immediately prior to dosing at multiple dosing (trough concentration) (Ctrough) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: AUCtau | Up to day 16
  AUC from the time of dosing to the start of the next dosing interval (AUCtau) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: Cmax | Up to day 16
  Maximum concentration (Cmax) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: PTR | Up to day 16
  Peak-trough ratio (PTR) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: Rac(AUC) | Up to day 16
  Accumulation ratio calculated using AUC (Rac(AUC)) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: Rac(Cmax) | Up to day 16
  Accumulation ratio calculated using Cmax (Rac(Cmax)) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: t1/2 | Up to day 16
  Terminal elimination half-life (t1/2) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: tmax | Up to day 16
  Time of the maximum concentration (tmax) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: MPR | Up to day 16
  Metabolite to parent ratio (MPR) will be recorded from the pharmacokinetic (PK) plasma samples collected.
Pharmacokinetics (PK) of ES259564 in plasma: Tlag | Up to day 16
  Time-lag (Tlag) will be recorded from the pharmacokinetic (PK) plasma samples collected.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma China, Inc.
Locations (1):
- Site CN86001, Bei'jing, China

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.